CLINICAL TRIAL: NCT06888973
Title: Mesenchymal Stem Cells Infusion in Patients With Autoimmune Diseases - A Phase II Clinical Trial
Brief Title: Mesenchymal Stem Cells Infusion in Patients With Autoimmune Diseases
Acronym: MSCs in AD
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Collaborators: Pak Emirates Military Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIBMT-MSC-autoimmune disease
Record Dates: First submitted 2025-01-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus (SLE); Systemic Sclerosis; Ankylosing Spondylitis (AS); Juvenile Idiopathic Arthritis; Polymyositis/Dermatomyositis
Keywords: Mesenchymal stem cells; Autoimmune diseases; Rheumatoid arthritis; Systemic Lupus Erythematosus (SLE); Systemic Sclerosis; Ankylosing Spondylitis (AS); Juvenile Idiopathic Arthritis; Polymyositis/dermatomyositis
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Spondylitis, Ankylosing; Arthritis, Juvenile; Dermatomyositis; Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Double-Blind, Randomized, Placebo-Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): MSC therapy group
  Interventions: Biological: Mesenchymal Stem Cells
- Placebo group (Placebo Comparator): Placebo (0.9% saline)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — allogeneic bone marrow-derived mesenchymal stem cells therapy
  Arms: Treatment group
Other: Placebo — 0.9% Saline as placebo
  Arms: Placebo group

SUMMARY:
The goal of this study is to learn if mesenchymal stem cell therapy (treatment group) can effectively treat autoimmune diseases, when compared to normal saline (given to placebo group). The primary outcome measures will be clinical improvement based on the respective disease specific clinical scores, normalization of T-lymphocyte subsets and > 50% reduction in disease specific antibody titres. The study will also document the type and frequency of any adverse event or side effects, reported by or seen in any of the trial participants.

Patients in treatment group will receive single session of MSC therapy and placebo group will receive 0.9% saline solution. The participants will be followed at 3 and 6 months.

DETAILED DESCRIPTION:
The autoimmune disorders are a spectrum of diseases ranging from organ-specific, in which antibodies and T cells react to self-antigens localized in a specific tissue, to systemic, which are characterized by reactivity against a specific antigen(s) spread throughout various tissues in the body. The incidence of different autoimmune diseases is variable, according to the Centers for Disease Control and Prevention, 22.7% have rheumatic diseases. Although no population-based epidemiological study has been carried out in Pakistan purely on autoimmune diseases; a study by Mohsin Z et al. reports the combined prevalence of rheumatic diseases at a tertiary hospital in Karachi to be 17.3%. Autoimmune diseases and their treatment modalities are the prime cause of disability in developing countries and have the highest incapacitating rates in health-related quality of life (HRQoL) and daily functioning.

The 21st century has seen rapid advances in the treatment of diseases of immune dysfunction. One such treatment modality is stem cell therapy which is believed to repair and regenerate tissues. In particular, mesenchymal stem cells (MSCs) have been applied to treat diseases associated with age, changing lifestyle, immune dysfunction and stroke. MSC therapy has promise to treat various autoimmune disorders like refractory systemic lupus erythematosus (SLE), Crohn's disease, systemic sclerosis (SS), rheumatoid arthritis (RA), multiple sclerosis (MS), graft versus host disease, diabetes mellitus, thyroiditis and even different types of neurological disorders. At present, nearly a thousand clinical trials have used MSC-based therapies. Among those around one hundred trials have been conducted for treatment of immune-mediated disorders, the first one being more than fifteen years ago (table 1).

The interest surrounding field of MSCs was initially based on their inherent capacity for self-renewal and regeneration with a potential to form cells of mesodermal origin (adipocytes, osteocytes, chondrocytes, hepatocytes, neurons, muscle cells and epithelial cells) depending on the surrounding microenvironment. Later on, due to their abilities to home to inflamed areas and exert immunomodulatory effects, therapies with MSCs extended to treatment of autoimmune and chronic inflammatory processes. Multiple studies have also demonstrated that MSCs have intrinsic immunomodulatory and anti-inflammatory properties.

Table 1: Clinical trials in which mesenchymal stem cells are being used as therapeutic modality.

Immune mediated disorder Number of Clinical trials Year of first Clinical trial Reference Graft vs. host disease 49 2004 Inflammatory bowel disease 23 2006 Multiple sclerosis 29 2006 Systemic lupus erythematosus 10 2007 Type I diabetes 26 2008 Primary Sjögren syndrome 1 2009 Type II diabetes 13 2010 Autoimmune hepatitis 2 2011 Ankylosing spondylitis 2 2011 Chronic urticarial 1 2017 Refractory autoimmune thrombocytopenia 1 2019

Source of MSCs MSCs were initially identified in the BM and are commonly isolated by gradient centrifugation to separate nucleated cells, followed by in vitro culture and serial passages. The Mesenchymal and Tissue Stem Cell Committee of the International Society for Cellular Therapy (ISCT) has designated the term 'multipotent mesenchymal stromal cells' for the plastic-adherent cells found under standard culture conditions. The immunophenotype of these cells as per ISCT criteria is positive for cell-surface markers CD73, CD90 and CD105 and negative for surface CD14 or CD11b, CD45, CD34, CD79 or CD19, and HLA-DR. MSCs have also been obtained from adipose tissue, placenta, amniotic fluid, umbilical cord blood (UCB), connective tissues of skeletal muscle and dermis,dental tissue, and fetal tissues such as lung and blood. Mobilized peripheral blood cells have also been reported as a source of MScs. Although gene expression studies demonstrate that MSC populations obtained from different tissue sources are highly heterogeneous, their ability to renew, differentiate, and major functional properties, such as regulation of immunological tolerance, wound healing, inflammation and fibrosis, are common to all MSCs.

1. Effects on cells of immune system MSCs suppress T-cell proliferation induced by alloantigens or mitogens via increasing the number of regulatory T cells and lessen complications of GVHD after HSCT and immune-mediated disease. In addition, MSCs inhibit function of B cells, natural killer cells and dendritic cells. The main immunosuppressive function of MSCs is by production of induced soluble factors; however, these cells can also exert immunosuppressive effects by direct cell-to-cell interaction. The immunosuppressive capacity of MSCs is enhanced under inflammatory conditions in the presence of the proinflammatory cytokines interferon (IFN)-g, tumor necrosis factor-alpha and interleukin (IL)-6.Under immunologically quiescent conditions, MSCs promote T-cell survival and can induce the activation and proliferation of CD4 positive regulatory T cells.
2. Production of immunomodulatory soluble factors MSCs constitutively produce inducible soluble factors, like transforming growth factor-β (TGF-β), hepatocyte growth factor, nitric oxide, HLA-G59 and indoleamine 2,3-dioxygenase that mediate their effects. Large amounts of IL-6 andIL-8, and the chemokine CCL-2 are also produced. MSCs treated with IFN-γ, secrete ICAM-1, CXCL-10 and CCL-8, whereas IL-8 production is decreased. This phenomenon suggests that MSCs target neutrophils and monocytes under non-inflammatory conditions, but attract monocytes, dendritic cells, T cells and natural killer cells under inflammatory conditions. A number of studies reported TGF-βas a key mediator of immunomodulation by MSCs.
3. Proinflammatory "licensing" of MSCs MSCs have been dubbed as ''smart" immune modulators since their suppressive effects require a previous licensing step that occurs in the presence of an inflammatory environment. If MSCs are transplanted during acute inflammation, the microenvironment containing polarized M1 macrophages 'licenses' MSCs to inhibit effector T, B, natural killer and dendritic cells. In contrast, if MSCs are licensed after the polarization of M2 macrophages by Th2-type cytokines as occurs during chronic inflammation, the microenvironment provides alternative licensing and recruits MSCs to the fibrosis process.
4. MSC paracrine factors in the repair mechanism Cellular regeneration of an ischemic tissue necessitates massive cell supply, on the order of a billion for an infarcted heart, for example. Experimental studies and clinical trials have revealed that MSC-mediated therapeutic benefit might largely rely on the contribution of the secreted amounts of growth factors and cytokines rather than on their potential for differentiation into cardiomyocytes, vascular or renal cells as shown by previous study. The panel of regulatory and trophic factors secreted by MSCs include a large number of growth factors, cytokines and chemokines.

Translation of MSC knowledge into clinical application Cell therapy indeed appears to be an applicable translational strategy for autoimmune diseases.

1. Graft versus Host Disease (GVHD) In humans, the most studied application for MSCs is GVHD, a complication of hematopoietic stem cell transplantation. In 2004, a 9-year-old boy with severe treatment-resistant acute GVHD of the gut and liver was treated with third-party haploidentical mother-derived MSCs. Phase II clinical trials in patients with steroid-resistant severe acute GVHD showed a 70% initial response rate that was not related to age or HLA match. However, durable complete responses or other primary endpoints in these trials are still lacking.
2. Crohn´s Disease (CD) The first report of a phase I clinical trial of cell therapy using autologous adipose-derived MSCs in CD was published in 2005. Local injection led to healing of fistulas (6/8) with no adverse effects These results were confirmed by the same group in 2009 in a phase II multicenter in a randomized controlled trial [24]. Currently, there is a phase III, multicenter, placebo-controlled, randomized and blind study to evaluate the safety and efficacy of allogeneic BM-MSCs, conducted by Osiris Therapeutics. (http://www.clinicaltrials. gov/ct2/show/NCT00482092).
3. Multiple Sclerosis (MS) Phase I/II studies in patients with refractory MS has confirmed the absence of adverse effects during follow-up (6-28 months). An increase in the proportion of CD4+CD25+ regulatory T cells with decreased proliferative responses of lymphocytes and activation markers on dendritic cells was detected hours after MSC transplantation. Patients improved on measures of visual function, without evidence of significant adverse events. Progression of general disability was also reduced after treatment.
4. Systemic Lupus Erythematosus (SLE) Perhaps the most remarkable results of human MSC therapy emerge now from clinical trials aimed at severe, treatment refractory SLE. Patients with active disease and lupus nephritis that was unresponsive to monthly i.v. cyclophosphamide and oral prednisone (≥ 20 mg/day) have shown improved outcomes when treated with MSCs. The Disease Activity Index (SLEDAI) in these patients improved significantly at one, six and twelve months follow-up, as did urinary protein. In some of the trials, patients with high SLEDAI received one infusion of allogeneic BM-MSCs from passage 3-5 from non HLA matched healthy family members. Their follow-up has reached a median of 17.2 (3-36) months, with no adverse effects, deaths or ensuing GVHD. Quite surprisingly, 24 h proteinuria decreased significantly as early as one week after MSC therapy, even preceding changes in anti-dsDNA antibodies, which decreased significantly at one month and three months post MSC dose. T regulatory (Treg) cells, found to be quantitatively and qualitatively deficient in active SLE, were restored at week one as judged by the percentage of CD4+ Foxp3+ cells among peripheral blood mononuclear cells. Other trials although with shorter follow-up also demonstrate significant improvement, verified for SLEDAI score, serum albumin, 24 h urinary protein, serum creatinine, serum complement and anti-dsDNA antibodies. Undoubtedly MSC therapy must be further explored in SLE.
5. Systemic Sclerosis (SS) SS is an immune mediated disease with a prominent vascular and microvascular component often leading to ischemic complications. Since MSCs can differentiate to endothelial cells in vitro and also participate in blood vessel formation in adult tissues, therapy both with autologous and haploidentical third party donor MSCs has been reported, leading to striking improvement in two separate case reports.
6. Rheumatoid Arthritis (RA) Literature search reveals that more than a hundred preclinical studies on RA animal model and nine clinical trials on human patients have been completed on use of MSC-based therapy in RA and establish its safety and efficacy. Whereas, nine clinical trials are still ongoing. In two-thirds of these patients a single dose of allogeneic MSCs at about a dose between 1-10 x106/kg were used. It is believed that MSCs targets the pathogenic memory T cells and halt the progression of disease course in RA patients.
7. Polymyositis/Dermatomyositis (PM/DM) Polymyositis/dermatomyositis (PM/DM) is an autoimmune disease characterized by weakness of proximal skeletal muscles and obvious skin manifestations, and is known to affect multiple organs, such as muscles, lungs, and kidneys. Currently, the etiology is not known. Several studies have suggested that T helper (Th) cells are involved in the pathogenesis of PM/DM, since Th cell-related cellular dysfunction plays an important role in the occurrence and development of PM or DM. Therefore, MSCT could provide a new therapeutic strategy for the treatment of PM and DM. Several studies have demonstrated that this approach has promising clinical outcomes. In another study 32 PM and DM patients were injected intravenously with 1 × 106/kg MSCs. The results of the 9-year follow-up study demonstrated that the symptoms and serological indicators of patients improved, showing the effectiveness and safety of MSCT in PM and DM, while 11 patients died due to reasons not related to transplantation.

In another study, 81 patients with PM/DM were randomly divided into two groups: 44 patients in the control group were individually treated with glucocorticoids and immunosuppressants for 6 months, while 37 patients in the transplantation group were injected intravenously with 3.5-5.2 × 107 UC-MSCs. The results of that study showed that the creatine kinase values in both groups were significantly decreased; however, the transplantation group had better results than the control group at several time points, and the lung function was significantly improved in the transplantation group. One patient died after transplantation and no transplantation-related complications occurred. Currently, there are only a few studies investigating PM/DM, and large-scale and randomized clinical studies are needed to evaluate the long-term effectiveness and safety of MSCT in PM/DM patients, including the risks of tumors and infections, as well as the optimal transplantation dose and schedule.

Since the clinical outcome in case reports and phase I-II trials seem occasionally striking, there exists a dire need to perform structured and preferably controlled multicenter trials and document results in our own population.

ELIGIBILITY:
Inclusion Criteria:

A- RA

* 18 Years and older
* Diagnosis of RA, as defined by fulfilling 2010 American College of Rheumatology (ACR) criteria
* Positive for rheumatoid factor (RF) and/or anticyclic citrullinated peptide (CCP)
* The presence of arthritis symptoms for more than 6 weeks but less than 5 year
* Active RA, as defined as DAS ESR>3.1 (as defined by moderate and sever RA )
* Willing to adhere to the study requirements
* Willing to use acceptable effective forms of contraception

Exclusion Criteria:

* • Allergy to methotrexate (MTX)

  * Previous exposure to anti-CD20 monoclonal antibody (mAb) or other type(s) of mAb therapy
  * Receipt of intra-articular injections within 4 weeks prior to study entry
  * Unwilling to stop drinking alcohol (ETOH)
  * History of alcohol or substance abuse
  * Active infection, or chronic or persistent infection that might worsen with immunosuppressive treatment (e.g., Human Immunodeficiency Virus [HIV], hepatitis B virus [HBV], hepatitis C virus [HCV], tuberculosis [TB])
  * Interstitial lung disease observed by chest x-ray [chest radiograph]
  * Known coronary artery disease or significant cardiac arrhythmias or severe congestive heart failure (New York Heart Association [NYHA] classes III or IV)
  * Definitive diagnosis of another autoimmune rheumatologic disease (e.g., systemic lupus erythematosus [SLE], scleroderma, primary Sjögren's syndrome, primary vasculitis)
  * History of immunoglobulin E (IgE)-mediated or non-IgE-mediated hypersensitivity or known anaphylaxis to mouse proteins
  * History of cancer. Exception: participants with previous resected basal or squamous cell carcinoma, treated cervical dysplasia, or treated in situ Grade I cervical cancer within 5 years prior to study entry are not excluded from study eligibility
  * History of positive purified protein derivative (PPD) test (i.e., positive tuberculosis [TB] test or mantoux test) without treatment for TB infection or chemoprophylaxis for TB exposure
  * Live vaccine within 3 months of study entry
  * Any psychiatric disorder that would prevent a participant from providing informed consent
  * Pregnancy or breastfeeding women.
  * HIV-positive patients.
  * Patients receiving any other investigational/disease modifying agents within 4 weeks of study entry.
  * History of allergic reactions attributed to compounds of similar biologic composition to mesenchymal stem cells.
  * Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent and perform all study assessments.
  * Active Malignancy
  * Any other serious medical illness that might preclude safe participation in the study.

Inclusion criteria for SLE

* Adults aged at least 18 years old
* Active musculoskeletal SLE diagnosed by SLICC criteria.
* No contraindication to the use of IV methylprednisolone, biosimilar rituximab, or any other required medications such as antipyretics and antihistamines
* Willing to use appropriate contraception if at risk of pregnancy
* Disease activity that is refractory to hydroxychoroquine and one DMARD, or patients unable to take hydroxychoroquine due to contra-indication or prior toxicity Exclusion criteria for SLE Severe "critical" SLE flare defined as: (i) BILAG 2004 A flare in CNS system; (ii) BILAG 2004 A flare in the renal system; or (iii) any other SLE manifestation requiring more immunosuppression than allowed within the protocol in the physician's opinion

  * Pregnancy
  * Breast Feeding
  * Malignancy
  * Receipt of intravenous immunoglobulin, plasma exchange or cyclophosphamide within the last 3 months
  * Rituximab within the past 18 months or other biologic therapies within the past 6 months
  * Active infections, including but not limited to the human immunodeficiency virus, hepatitis B (including prior infection as judged by positive Hepatitis B core antibody) or hepatitis C
  * Receipt of a live attenuated vaccine within 3 months prior to study enrolment
  * History of cancer in the past 5 years except for squamous or basal cell carcinoma that has been completely excised or treated cervical carcinoma in situ
  * Planned surgery within the study period that is expected to require overnight hospital admission
  * Any other concomitant medical condition that, in the investigator's opinion, or after discussion with the CI, places the participant at risk by participating in this study Inclusion criteria for systemic sclerosis
* Adult patients, >/= 18 years of age
* Systemic sclerosis, as defined by American College of Rheumatology (1980) criteria
* Disease duration upto 5 years (defined as time from first non-Raynaud phenomenon manifestation)
* >/= 15 and </= 40 mRSS units at screening
* Active disease, as defined by protocol
* Negative pregnancy test for a female subject of childbearing potential Exclusion criteria
* Major surgery (including joint surgery) within 8 weeks prior to and/or during study enrollment
* Rheumatic autoimmune disease other than systemic sclerosis
* Previous treatment with tocilizumab
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Severe cardiopulmonary disease
* Known active current or history of recurrent infections
* Use of any investigational, biologic, or immunosuppressive therapies .
* Primary or secondary immunodeficiency Inclusion criteria for ankylosing spondlitis Male or non-pregnant, non-lactating female patients at least 18 years of age

Diagnosis of moderate to severe AS with prior documented radiologic evidence (x-ray or radiologist's report) fulfilling the Modified New York criteria for AS:

* Active AS assessed by BASDAI ≥4 (0-10) at Baseline
* Spinal pain as measured by BASDAI question #2 ≥ 4 cm (0-10 cm) at Baseline
* Total back pain as measured by VAS ≥ 40 mm (0-100 mm) at Baseline Patients should have had inadequate response or failure to respond to at least 2 NSAIDs at an approved dose for a minimum of 4 weeks in total and a minimum of 2 weeks for each NSAID prior to randomization, or less than 4 weeks if therapy had to be withdrawn due to intolerance, toxicity or contraindications Patients who are regularly taking NSAIDs (including COX-1 or COX-2 inhibitors) as part of their AS therapy are required to be on a stable dose for at least 2 weeks before randomization patients who have been on a TNFα inhibitor (not more than one) must have experienced an inadequate response to previous or current treatment given at an approved dose for at least 3 months prior to randomization or have been intolerant to at least one administration of an anti-TNFα agent Exclusion criteria for ankylosing spondlitis

  * Chest X-ray or MRI with evidence of ongoing infectious or malignant process
  * Previous exposure to secukinumab or any other biologic drug directly targeting IL-17 or IL-17 receptor
  * Pregnant or nursing (lactating) women Inclusion criteria for dermatomyositis
* 5 to 50 Years of age
* Adults with definite or probable dermatomyositis or polymyositis and pediatric patients five years of age and over with definite or probable juvenile dermatomyositis by Bohan and Peter criteria. Diagnosis of JDM based on an age of onset (i.e., first symptom of myositis or dermatomyositis rash) is less 16 years of age
* Refractory myositis, defined by intolerance to or inadequate response to corticosteroids plus an adequate regime of at least one other immunosuppressive agent. Intolerance is defined as side effects that require discontinuation of the medication or an underlying condition that precludes further use of the medication.
* Baseline manual muscle testing which is based on a maximum MMT-8 (Manual Muscle Test) score of 150:Adult subjects with dermatomyositis (DM) or polymyositis (PM) must have a score that is no greater than 125/150 in conjunction with 2 other abnormal core set measures.

Subjects with a diagnosis of Juvenile Dermatomyositis (JDM) must meet either of the following criteria:

1. An MMT-8 (Manual Muscle Test) score that is no greater than 125/150 in conjunction with 2 other abnormal core set measures.

   OR
2. If MMT (Manual Muscle Test) score is greater than 125/150 the patient MUST meet at least 3 abnormal core set measures.

   * Background therapy with at least 1 non-corticosteroid immunosuppressive agent at a stable dose for at least 6 weeks prior to screening
   * Able and willing to complete self-report questionnaires. Parents of pediatric participants will be required to complete the questionnaires on behalf of their children.
   * Willing to use acceptable forms of contraception for the duration of the study for patients of reproductive potential.
   * Parent willing to provide informed consent, if applicable
   * Willing to forgo immunization with a live vaccine for the duration of the study Exclusion for dermatomyositis

     * Drug-induced myositis. Patients who have myositis or myopathic syndromes caused by taking medications known to induce myositis-like syndromes, including but not limited to statin agents, fibric acid derivatives, colchicine, and hydroxychloroquine.
     * Inclusion body myositis
     * Cancer-associated myositis, defined as the diagnosis of myositis within 2 years of the diagnosis of cancer. Patients with basal or squamous cell skin cancer or carcinoma in situ of the cervix are not excluded, if it has been at least 5 years since excision.
     * Myositis in overlap with another connective tissue disease that may preclude the accurate assessment of a treatment response
     * Live viral vaccine within 4 weeks prior to study entry
     * Any joint disease or other musculoskeletal condition that may interfere with muscle strength testing
     * Known hypersensitivity to mouse proteins
     * Any concomitant or life-threatening non-myositis illness that, in the opinion of the investigator, may interfere with the study
     * Known or suspected history of drug or alcohol abuse within the last 6 months prior to study entry, as determined by medical record or patient interview
     * Anticipated poor compliance with study requirements
     * Participation in another clinical trial within 30 days prior to screening
     * Any history or evidence of any severe illness or other condition that, in the opinion of the investigator, may interfere with the study
     * Previously received rituximab
     * Evidence of prior infection with hepatitis B or hepatitis C virus
     * Initiation of an exercise program within 4 weeks of screening OR initiation of an exercise program during the study
     * Consumed any creatine-containing, over-the-counter products in the form of dietary supplements 30 days prior to screening visit and for the duration of the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in the Disease Activity Score- Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 48 The DAS28-ESR is a score on a scale (0 to 10) that is a measure of the subject's disease activity. It is based on the tender joint count (28 joints), swollen joint count (28 joints), patient's global assessment of disease activity (mm), and ESR (mm/hour). Lower score indicates less disease activity. Flares in disease activity are defined as an increase in this score of greater than 1.2 and remission is defined as achieving a DAS28-ESR score of less than 2.6.
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Tender Joint Count Score at Week 48 Tender Joint Count (TJC) is calculated based on tenderness response of 28 joints. TJC possible values range from 0 to 28. A lower TJC indicates less joint tenderness. Change from baseline is computed as Week 48 value minus baseline value. A negative value in change from baseline indicates an improvement.
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Swollen Joint Count at Week 48 Swollen Joint Count (SJC) is calculated based on swelling response of 28 joints. SJC possible values range from 0 to 28. A lower SJC indicates less joint swelling. Change from baseline is computed as Week 48 value minus baseline value. A negative value in change from baseline indicates an improvement
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Patient's Assessment of Arthritis Pain-Visual Analog Scale (PAAP-VAS) at Week 48 Change from Baseline in PAAP-VAS (0 to 100 millimeters visual analog scale, 0 being no pain and 100 being most severe pain) is computed as the value at Week 48 minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Patient's Global Assessment of Disease Activity- Visual Analog Scale (PtGADA-VAS) at Week 48 Change from Baseline in PtGADA-VAS (0 to 100 mm visual analog scale, 0 being no symptoms and 100 being severe symptoms) is computed as the value at Week 48 minus the Baseline value. A negative value in change from Baseline indicates an improvement.
Primary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Physician's Global Assessment of Patient's Disease Activity- Visual Analog Scale (PhGADA-VAS) at Week 48
Primary Outcome Measures for Systemic lupus erythematosus | Day 0, Weeks 12, 24, 48
  Proportion of patients achieving BILAG-based Composite Lupus Assessment (BICLA)
Primary Outcome Measures for systemic sclerosis | Day 0, Weeks 12, 24, 48
  Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 48 Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement.
Primary Outcome Measures for systemic sclerosis | Day 0, Weeks 12, 24, 48
  Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Primary outcome measures in ankylosing spondlitis | Week 16
  The Proportion of Participants Who Achieve an ASAS 20 Response (Assessment of SpondyloArthritis International Society Criteria) ASAS20 response is defined as an improvement of ≥20% and ≥1 units on a scale of 10 in at least three of the four ASAS main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain
Primary Outcome Measure for dermatomyositis | Day 0, Weeks 12, 24, 48
  Comparison Between the Time to Improvement Between the Two Groups of Idiopathic Inflammatory Myopathy Patients at week 48 ASAS20 response is defined as an improvement of ≥20% and ≥1 units on a scale of 10 in at least three of the four ASAS main domains and no worsening of ≥20% and ≥1 unit on a scale of 10 in the remaining domain

SECONDARY OUTCOMES:
Secondary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in the Short Form 36 (SF-36) Physical and Mental Health Component Summary Scores (PCS and MCS) at Week 48 [ Time Frame: Baseline (Day 0), Week 12,week 24,week48 ] It has 36 questions with 8 subscale scores and 2 summary scores: PCS=physical functioning, role-physical, bodily pain, and general health; MCS=vitality, social functioning, role-emotional, and mental health. Scoring is done for both subscores and summary scores. For both, 0=worst score (or quality of life) and 100=best score. Change from baseline is computed as the value at Week 48 minus the baseline value. A positive value in change from Baseline indicates an improvement and a negative value worsening.
Secondary Outcome Measures for RA | Day 0, Weeks 12, 24, 48
  Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 48 [ Time Frame:
  Each question is scored 0-3 (0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do). In addition, category scores are modified if an aid or device is used, for example, a walker or wheelchair, or help is received from another person in the daily living activities. If an aid or device is used or help is received then a category score of 0 or 1 increases to a category score of 2. A category score of 3 remains a 3 regardless of aids, devices, or help. Scores from each of the 8 categories are totaled. The total score can range from 0 to 24. Change from baseline is computed as the total score at Week 48 minus the baseline total score. A negative value in change from baseline indicates an improvement.
Secondary Outcome Measures for RA | Day 0, Week 12, week 24, week48
  Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Week 48 ESR is a blood test used to monitor therapy in inflammatory diseases such as rheumatoid arthritis and reflects acute phase reactant levels. Active disease in RA is defined by an ESR greater than 30 mm/hr. Change from baseline is computed as the value at Week 48 minus the baseline value. A negative value in change from baseline indicates an improvement
Secondary Outcome Measures for SLE | Day 0, Weeks 12, 24, 48
  Proportion of patients achieving SLEDAI responder Index (SRI)
Secondary Outcome Measures for SLE | Day 0, Weeks 12, 24, 48
  Number of serious adverse events
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Physical Function Assessed by Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI) Each VAS item was rated separately (0-100 millimeters [mm]), with higher scores indicating more severe disease. The five items were: 1) intestinal disease, 2) breathing problem, 3) Raynaud syndrome, 4) finger ulcers, and 5) overall disease.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) There are four possible responses for each component: 0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty; 3 = unable to do. The HAQ-DI was the sum of the domain scores, divided by the number of domains that have a score (i.e. the average score), with total range of 0 to 3, higher scores showing larger functional limitation.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Clinician's Global Assessment The Clinician's Global Assessment evaluated the overall impact of SSc on the participant as assessed by the physician on a VAS with scores ranging from 0 to 100 mm, with higher scores indicating worse disease in terms of severity, damage, or overall disease, but there was no standardization for the scale.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Patient's Global Assessment VAS scale (0 mm to 100 mm), with higher scores indicating worsening disease.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score The endpoint measured was fatigue. On this scale, a numerical increase indicated an improvement in the participant's condition.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in 5-D Itch Scale Each domain was scored on a 5-point scale, the scores of each of the five domains were achieved separately and then summed together to obtain a total 5-D score. 5-D scores ranged between 5 (no pruritus) and 25 (most severe pruritus).
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in mRSS
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Percentage of Participants who maintained or Improved in mRSS
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Change From Baseline in Tender Joint Count 10 proximal interphalangeal joint (PIP) joints, and both knees, were assessed. Joints were classified as not tender = 0 or tender = 1. Observed data was presented for this outcome measure.
Secondary Outcome Measures for SC | Day 0, Weeks 12, 24, 48
  Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Secondary Outcome Measure for ALS | Week 16
  The Proportion of Participants Who Achieve an ASAS40 Response ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 10 in at least three of the four ASAS main domains and no worsening at all in the remaining domain
Secondary Outcome Measure for ALS | Week 16
  The Proportion of Participants Who Achieve an ASAS40 Response
Secondary Outcome Measure for ALS | Week 16
  Change in high-sensitivity C-reactive protein (hsCRP) Over Time
Secondary Outcome Measure for ALS | Week 16
  Percentage of Participants Who Achieve an ASAS 5/6 The ASAS 5/6 improvement criteria is an improvement of ≥20% in at least five of all six domains
Secondary Outcome Measure for ALS | Week 16
  Participants With Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Response The BASDAI or Bath Ankylosing Spondylitis Disease Activity Index consists of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which is used to answer 6 questions pertaining to the 5 major symptoms of AS
Secondary Outcome Measure for ALS | Week 16
  Change in Short Form (36) Physical Component Summary (PCS) Responders (Improvement of >= 2.5 Points) at Week 16
Secondary Outcome Measure for ALS | Week 16
  Change in Ankylosing Spondylitis Quality of Life (ASQoL) Score Over Time The Ankylosing Spondylitis Quality of Life (ASQoL) is an instrument to assess health-related quality of life among adult patients with Ankylosing Spondylitis.
  Each statement on the ASQoL is given a score of "1" or "0". A score of "1" is given where the item is affirmed, indicating adverse QoL. All item scores are summed to give a total score or index. Scores can range from 0 (good QoL) to 18 (poor QoL).
Secondary Outcome Measure for ankylosing spondlitis | Week 16
  The Proportion of Patients Who Achieve an The Assessment in SpondyloArthritis International Society (ASAS) Partial Remission The The Assessment in SpondyloArthritis International Society (ASAS) partial remission criteria are defined as a value not above 2 units in each of the four main domains on a scale of 10
Secondary Outcome Measure for dermatomyositis | Day 0, Weeks 12, 24, 48
  Response Rates (Proportion of Improved Patients) The Definition of Improvement for both adult and pediatric patients will be: 3 of any of the 6 core set measures improved by ≥ 20%, with no more than 2 of the core set measures worsening by ≥25% (worsening measure cannot include the MMT) at two consecutive visits. Of note, the MMT could not be one of the worsening measures.
Secondary Outcome Measure for dermatomyositis | Day 0, Weeks 12, 24, 48
  20% Improvement in Manual Muscle Testing (MMT) Over Baseline on Two Consecutive Time Points (Muscle is the Primary Organ of Involvement, and MMT is the One Objective Measurement of the Definition of Improvement [DOI])

CONTACTS AND LOCATIONS:
Overall Officials: Memoona Haider, MBBS, FCPS, Study Chair — National University of Medical Sciences
Locations (2):
- Pakistan (2):
  - Armed Forces Bone Marrow Transplant Centre/ National Institute of Blood and Marrow Transplant (AFBMTC/NIBMT), Rawalpindi
  - Pak Emirates Military Hospital, Rawalpindi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Blanc K, Frassoni F, Ball L, Locatelli F, Roelofs H, Lewis I, Lanino E, Sundberg B, Bernardo ME, Remberger M, Dini G, Egeler RM, Bacigalupo A, Fibbe W, Ringden O; Developmental Committee of the European Group for Blood and Marrow Transplantation. Mesenchymal stem cells for treatment of steroid-resistant, severe, acute graft-versus-host disease: a phase II study. Lancet. 2008 May 10;371(9624):1579-86. doi: 10.1016/S0140-6736(08)60690-X. PMID 18468541
- [Background] Laflamme MA, Murry CE. Regenerating the heart. Nat Biotechnol. 2005 Jul;23(7):845-56. doi: 10.1038/nbt1117. PMID 16003373
- [Background] Viswanathan S, Shi Y, Galipeau J, Krampera M, Leblanc K, Martin I, Nolta J, Phinney DG, Sensebe L. Mesenchymal stem versus stromal cells: International Society for Cell & Gene Therapy (ISCT(R)) Mesenchymal Stromal Cell committee position statement on nomenclature. Cytotherapy. 2019 Oct;21(10):1019-1024. doi: 10.1016/j.jcyt.2019.08.002. Epub 2019 Sep 13. PMID 31526643
- [Background] Choi YH, Kurtz A, Stamm C. Mesenchymal stem cells for cardiac cell therapy. Hum Gene Ther. 2011 Jan;22(1):3-17. doi: 10.1089/hum.2010.211. PMID 21062128
- [Background] Nauta AJ, Fibbe WE. Immunomodulatory properties of mesenchymal stromal cells. Blood. 2007 Nov 15;110(10):3499-506. doi: 10.1182/blood-2007-02-069716. Epub 2007 Jul 30. PMID 17664353
- [Background] Lee OK, Kuo TK, Chen WM, Lee KD, Hsieh SL, Chen TH. Isolation of multipotent mesenchymal stem cells from umbilical cord blood. Blood. 2004 Mar 1;103(5):1669-75. doi: 10.1182/blood-2003-05-1670. Epub 2003 Oct 23. PMID 14576065
- [Background] Owen M, Friedenstein AJ. Stromal stem cells: marrow-derived osteogenic precursors. Ciba Found Symp. 1988;136:42-60. doi: 10.1002/9780470513637.ch4. PMID 3068016
- [Background] Kabat M, Bobkov I, Kumar S, Grumet M. Trends in mesenchymal stem cell clinical trials 2004-2018: Is efficacy optimal in a narrow dose range? Stem Cells Transl Med. 2020 Jan;9(1):17-27. doi: 10.1002/sctm.19-0202. Epub 2019 Dec 5. PMID 31804767
- [Background] Mizuno H. Adipose-derived stem cells for tissue repair and regeneration: ten years of research and a literature review. J Nippon Med Sch. 2009 Apr;76(2):56-66. doi: 10.1272/jnms.76.56. PMID 19443990
- [Background] Song H, Song BW, Cha MJ, Choi IG, Hwang KC. Modification of mesenchymal stem cells for cardiac regeneration. Expert Opin Biol Ther. 2010 Mar;10(3):309-19. doi: 10.1517/14712590903455997. PMID 20132054
- [Background] Phinney DG, Prockop DJ. Concise review: mesenchymal stem/multipotent stromal cells: the state of transdifferentiation and modes of tissue repair--current views. Stem Cells. 2007 Nov;25(11):2896-902. doi: 10.1634/stemcells.2007-0637. Epub 2007 Sep 27. PMID 17901396
- [Background] Choi EW, Shin IS, Lee HW, Park SY, Park JH, Nam MH, Kim JS, Woo SK, Yoon EJ, Kang SK, Ra JC, Youn HY, Hong SH. Transplantation of CTLA4Ig gene-transduced adipose tissue-derived mesenchymal stem cells reduces inflammatory immune response and improves Th1/Th2 balance in experimental autoimmune thyroiditis. J Gene Med. 2011 Jan;13(1):3-16. doi: 10.1002/jgm.1531. PMID 21259404
- [Background] Cai L, Johnstone BH, Cook TG, Tan J, Fishbein MC, Chen PS, March KL. IFATS collection: Human adipose tissue-derived stem cells induce angiogenesis and nerve sprouting following myocardial infarction, in conjunction with potent preservation of cardiac function. Stem Cells. 2009 Jan;27(1):230-7. doi: 10.1634/stemcells.2008-0273. PMID 18772313
- [Background] Augello A, Tasso R, Negrini SM, Cancedda R, Pennesi G. Cell therapy using allogeneic bone marrow mesenchymal stem cells prevents tissue damage in collagen-induced arthritis. Arthritis Rheum. 2007 Apr;56(4):1175-86. doi: 10.1002/art.22511. PMID 17393437
- [Background] Zappia E, Casazza S, Pedemonte E, Benvenuto F, Bonanni I, Gerdoni E, Giunti D, Ceravolo A, Cazzanti F, Frassoni F, Mancardi G, Uccelli A. Mesenchymal stem cells ameliorate experimental autoimmune encephalomyelitis inducing T-cell anergy. Blood. 2005 Sep 1;106(5):1755-61. doi: 10.1182/blood-2005-04-1496. Epub 2005 May 19. PMID 15905186
- [Background] Yanez R, Lamana ML, Garcia-Castro J, Colmenero I, Ramirez M, Bueren JA. Adipose tissue-derived mesenchymal stem cells have in vivo immunosuppressive properties applicable for the control of the graft-versus-host disease. Stem Cells. 2006 Nov;24(11):2582-91. doi: 10.1634/stemcells.2006-0228. Epub 2006 Jul 27. PMID 16873762
- [Background] Garcia-Gomez I, Elvira G, Zapata AG, Lamana ML, Ramirez M, Castro JG, Arranz MG, Vicente A, Bueren J, Garcia-Olmo D. Mesenchymal stem cells: biological properties and clinical applications. Expert Opin Biol Ther. 2010 Oct;10(10):1453-68. doi: 10.1517/14712598.2010.519333. PMID 20831449
- [Background] Parekkadan B, Milwid JM. Mesenchymal stem cells as therapeutics. Annu Rev Biomed Eng. 2010 Aug 15;12:87-117. doi: 10.1146/annurev-bioeng-070909-105309. PMID 20415588
- [Background] Si YL, Zhao YL, Hao HJ, Fu XB, Han WD. MSCs: Biological characteristics, clinical applications and their outstanding concerns. Ageing Res Rev. 2011 Jan;10(1):93-103. doi: 10.1016/j.arr.2010.08.005. Epub 2010 Aug 19. PMID 20727988
- [Background] Mohsin Z, Asghar AA, Faiq A, Khalid I, Ul-Haque I, Rehman S, Ahmed SI, Basalat ST, Aimen A, Shafique S, Hanif A, Iqbal MW, Samad SA, Siddiqui F, Hameed I, Safri M. Prevalence of Rheumatic Diseases in a Tertiary Care Hospital of Karachi. Cureus. 2018 Jun 22;10(6):e2858. doi: 10.7759/cureus.2858. PMID 30148011
- [Background] Cooper GS, Stroehla BC. The epidemiology of autoimmune diseases. Autoimmun Rev. 2003 May;2(3):119-25. doi: 10.1016/s1568-9972(03)00006-5. PMID 12848952